CLINICAL TRIAL: NCT03704753
Title: New Truncal Nerve Blocks for Thoracoscopic Surgery and Open Heart Surgery.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tampere University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R18011M
Record Dates: First submitted 2018-10-10; First posted 2018-10-15 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2022-10

CONDITIONS: Postoperative Pain
Keywords: Cardiac Surgery; Thoracic Surgery; Nerve block
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Randomised and double blinded.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- SAPB group A (Active Comparator): SAPB single injection. 30ml of Ropivacaine 7,5mg/ml is injected above m. serratus anterior after thoracoscopic lung surgery. Infection is done under ultrasound guidance.
  Interventions: Drug: Ropivacaine
- SAPB group B (Placebo Comparator): SAPB single injection (placebo). 30ml of SodiumChloride 0.9 is injected above m. serratus anterior after thoracoscopic lung surgery. Infection is done under ultrasound guidance.
  Interventions: Drug: Sodium chloride 0.9%
- SAPB group C (Active Comparator): SAPB single injection and catheter. 30ml of Ropivacaine 7,5mg/ml is injected above m. serratus anterior after thoracoscopic lung surgery and a multi-holed catheter is left in place. 20ml of Ropivacaine 2mg/ml is injected every 12h through catheter postoperatively.
  Interventions: Drug: Ropivacaine
- SAPB group D (Active Comparator): Continious intercostal catheter. 20ml of Ropivacaine 7,5mg/ml is injected through intercostal catheter, which i placed under thoracoscopic visualization. After single injection a continuous infusion of Ropivacaine 2mg/ml is started (weight dependent daily dosage).
  Interventions: Drug: Ropivacaine
- SIP group A (Active Comparator): SIP single injection 20ml of Ropivacaine 7,5mg/ml is injected under pectoralis major muscle on both sides of sternum. Injection is done under ultrasound guidance.
  Interventions: Drug: Ropivacaine
- SIP group B (Placebo Comparator): SIP single injection (placebo) 20ml of SodiumChloride 0.9 is injected under pectoralis major muscle on both sides of sternum. Injection is done under ultrasound guidance.
  Interventions: Drug: Sodium chloride 0.9%

INTERVENTIONS:
Drug: Ropivacaine — Serratus anterior plane block for thoracic surgery patients and subpectoral interfascial nerve block for open heart surgery patients
  Arms: SAPB group A; SAPB group C; SAPB group D; SIP group A
Drug: Sodium chloride 0.9% — Serratus anterior plane block for thoracic surgery patients and subpectoral interfascial nerve block for open heart surgery patients (placebo).
  Arms: SAPB group B; SIP group B

SUMMARY:
This study is divided to two sub-studies. First sub-study evaluates if Serratus Anterior Plane block (SAPB) reduces opioid consumption after thoracoscopic surgery. Secondly continuous SAPB is compared to continuous intercostal blockade. Second sub-study evaluates if Subpectoral Interfascial Plane block (SIP) reduces opioid consumption after medial sternotomy.

DETAILED DESCRIPTION:
Serratus anterior plane block (SAPB) - sub-study

In this sub-study 120 patients will be randomly assigned to one of four groups:

SAPB group A 30ml of Ropivacaine 7,5mg/ml is injected above m. serratus anterior after thoracoscopic lung surgery. Injection is done under ultrasound guidance.

SAPB group B 30ml of Sodiumchloride 0.9 is injected above m. serratus anterior after thoracoscopic lung surgery. Injection is done under ultrasound guidance.

SAPB group C 30ml of Ropivacaine 7,5mg/m is injected above m. serratus anterior after thoracoscopic lung surgery. Also a multi-holed catheter is left in place. Through catheter 20ml Ropivacaine 2mg/ml is injected every 12 hours after surgery.

SAPB group D A multi-holed catheter is placed in single intercostal space under thoracoscopic visualization. 20ml of Ropivacaine 7,5mg/ml is injected after application of the catheter, also a continuous infusion of ropivacaine 2mg/ml is started. Rate of the infusion is determined by patients weight.

Subpectoral Interfascial Plane block (SIP) - sub-study

In this sub-study 80 patients will be randomly assigned to one of two groups:

SIP group A 20ml of ropivacaine 7,5mg/ml is injected under both pectoralis major muscles before medial sternotomy. Injection is done under ultrasound guidance.

SIP group B 20ml of sodiumchloride 0.9 is injected under both pectoralis major muscles before medial sternotomy. Injection is done under ultrasound guidance.

Every patients postoperative pain is treated with intravenous oxycodone PCA-pump.

The investigators will evaluate post operative pain based on the Numeric rating Scale, 24 hours oxycodone consumption. The investigators will also evaluate post operative chronic pain using three questionnaires: EQ5D, STAIT-TRAIT and Pain Detect. In SAPB sub-study the questionnaires are done three weeks and 6 months post. operatively. In SIP sub-study the questionnaires are done 6 months and 12 months post.operatively.

ELIGIBILITY:
Inclusion Criteria:

* Elective thoracoscopic lung surgery or elective open heart valve surgery

Exclusion Criteria:

* DM1 with complications, lack of co-operation, refusal, chronic pain, chronic intake of opioids or use of SNRI or tricyclic antidepressants.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-01-25 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Opioid consumption | 24 postoperative hours
  Oxycodone

CONTACTS AND LOCATIONS:
Locations (1):
- Tampere Heart Hospital, Tampere, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kalli A, Vistbacka J, Moilanen E, Jarvela K, Mennander A. Superficial Parasternal Intercostal Plane Block and Full Sternotomy; A Randomized Trial. Eur J Cardiothorac Surg. 2025 Jul 1;67(7):ezaf226. doi: 10.1093/ejcts/ezaf226. PMID 40627369